CLINICAL TRIAL: NCT05558111
Title: Neuroimaging Study of Supraspinal Control of Lower Urinary Tract Function in Patients with Orthotopic Sigmoid Neobladder.
Brief Title: The Supraspinal Control of Lower Urinary Tract Function in Patients with Orthotopic Sigmoid Neobladder.
Status: Recruiting | Type: Observational
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Principal Investigator, Chunxiao Liu, Professor;Chief Surgeon, Zhujiang Hospital
Other Study IDs: 2022-KY-131-02
Record Dates: First submitted 2022-09-24; First posted 2022-09-28 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-09

CONDITIONS: Orthotopic Neobladder
Keywords: Orthotopic neobladder; Functional magnetic resonance imaging; Neuroimaging Study; Lower urinary tract function; Bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with orthotopic neobladder: Patients with orthotopic neobladder who met the inclusion criteria will be enrolled.Inclusion criteria :(1) being right-handed;(2) 3 months or more after operation;(3) No contraindications to fMIR examination;(4)Does not meet the relevant exclusion criteria.

SUMMARY:
Orthotopic sigmoid neobladder surgery is one of the ideal urinary diversion methods after radical cystectomy.In recent years, functional imaging studies have revealed brain regions related to urinary system function, but brain activity of lower urinary tract function in neobladder patients is still unclear.The aim of this study is to explore the brain activity of urination intention and self-controlled urination behavior in patients with orthotopic sigmoid neobladder by task-state functional magnetic resonance imaging (fMRI).

ELIGIBILITY:
Inclusion Criteria:

1. Being right-handed;
2. 3 months or more after operation;
3. No contraindications to fMIR examination;
4. Voluntarily sign informed consent.

Exclusion Criteria:

1. History of bladder radiotherapy;
2. History of prostate cancer;
3. Suffering from diseases affecting abdominal pressure;
4. History of abnormal brain anatomy, craniocerebral surgery, craniocerebral tumor, and craniocerebral radiotherapy;
5. History of mental disorders, Parkinson's disease, Alzheimer's disease, epilepsy, cerebral infarction, cerebral hemorrhage;
6. Claustrophobia or carrying metal implants that are not suitable for fMRI examination;
7. Diseases affecting lower urinary tract function (such as spinal cord injury, diabetic peripheral neuropathy, etc.);
8. Urethral stricture;
9. Refusing to sign the informed consent form for clinical projects;
10. Other conditions that were not suitable for inclusion according to the investigator's judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients 3 months or more after orthotopic neobladder surgery.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
The location of brain functional activation areas | 3 months
  Areas of the brain where excitation or inhibition occurs in fMRI images
The peak T-value size of the activation region | 3 months
  Peak T values of activated or inhibited regions of the brain in fMRI images

CONTACTS AND LOCATIONS:
Overall Officials: Chunxiao Liu, Principal Investigator — Southern Medical University, China
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China